CLINICAL TRIAL: NCT06426420
Title: Detection of Endometriosis Using ATR-FTIR Spectroscopy
Brief Title: Endometriosis and ATR-FTIR Spectroscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Espirito Santo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, VALERIO GARRONE BARAUNA, Professor, Federal University of Espirito Santo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FTIR-ENDOMETRIOSIS
Record Dates: First submitted 2024-05-14; First posted 2024-05-23 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Endometriosis; Endometriomas
Keywords: Endometriosis; Diagnosis; Spectroscopy; FTIR; Urine; Detection; Infrared
MeSH Terms: conditions — Endometriosis; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pelvic Pain (Experimental): Patients referred to the gynecology outpatient clinic, with complain of pelvic pain. Positives and negatives for endometriosis will be outlined by an expert gynecologist according to the following criteria:
  * Pelvic MRI (Magnetic Resonance Imaging) report;
  * Gynecologic exam;
  * Clinical symptoms and history;
  The intervention is the use of the ATR-FTIR Spectrometer in patient's urine samples to develop and validate a tool for detecting endometriosis.
  Interventions: Diagnostic Test: FTIR spectroscopy analysis

INTERVENTIONS:
Diagnostic Test: FTIR spectroscopy analysis — ATR-FTIR Spectroscopy analysis combined with machine learning algorithms.

SUMMARY:
The goal of this study is to explore the use of mid-infrared spectroscopy (ATR-FTIR) as a detection tool for endometriosis in urine.

DETAILED DESCRIPTION:
Endometriosis is a chronic gynecological disease that is considered debilitating and multifactorial. Its diagnosis is invasive and can be prolonged due to non-specific symptoms and erroneous or late investigations, which can lead to delays and impair the provision of adequate treatment.

ATR-FTIR Spectroscopy is a non-invasive technique with the capability to identify the chemical composition and molecular changes of samples through its interaction with mid-infrared radiation. The aim of this work is to develop a rapid test for the detection of endometriosis in urine samples using spectroscopy and machine learning algorithms.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Pelvic pain complain

Exclusion Criteria:

* Age under 18 or above 55
* Lack of informed consent

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Biological woman self-identified as woman
Enrollment: 600 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2026-04-29 (Estimated); Study Completion 2026-04-29 (Estimated)

PRIMARY OUTCOMES:
Spectroscopy Reliability (diagnostic metrics) | 1 year
  The primary outcome is the evaluation of specificity, sensitivity and accuracy of the diagnostic. Acceptable diagnostic metrics must be comparable to MRI, which will demonstrate if spectroscopy can discriminate between negative and positive endometriosis patients.

CONTACTS AND LOCATIONS:
Overall Officials: Valerio G Barauna, PhD, Principal Investigator — Universidade Federal do Espírito Santo
Locations (1):
- University Hospital Cassiano Antonio Moraes at Federal Univeristy Of Espírito Santo, Vitória, Espírito Santo, Brazil

IPD SHARING:
Plan to Share IPD: No